CLINICAL TRIAL: NCT01387503
Title: Controlled Expansion of Conventional Criteria for Liver Transplantation in Hepatocellular Carcinoma Through Downstaging Procedures: a Randomized Trial (XXL Trial)
Brief Title: Expansion of Conventional Criteria for Liver Transplantation in Hepatocellular Carcinoma Through Downstaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: AISF (Associazione Italiana per lo Studio del Fegato) (Unknown); CNT (Centro Nazionale Trapianti) (Unknown); NITp (Nord Italia Transplant project) (Unknown); OCST (Organizzazione Centro Sud Trapianti) (Unknown); Associazione Italiana per la Ricerca sul Cancro (Other); Ministero della Salute, Italy (Other); Basilicata Region (Unknown)
Responsible Party: Principal Investigator, Vincenzo Mazzaferro, Professor, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INT 80/09
Record Dates: First submitted 2011-06-30; First posted 2011-07-04 (Estimated); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Carcinoma, Hepatocellular; Cirrhosis
Keywords: Hepatocellular Carcinoma; Liver Transplantation; Downstaging; Trans-arterial chemoembolization (TACE); Radiofrequency ablation (RFA); Liver resection; Sorafenib
MeSH Terms: conditions — Carcinoma, Hepatocellular; Fibrosis | interventions — Liver Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 - Transplant strategy (Experimental): Patients randomized to Group 1 will be enlisted for liver transplantation and will undergo liver transplantation within 8 months unless oncological (i.e. extrahepatic disease) or medical (i.e. cardiac insufficiency) will occur
  Interventions: Procedure: Liver transplantation
- Group 2 - Non-transplant strategy (No Intervention): Patients randomized to Group 2 will continue to receive treatments according to their stage of disease, or will undergo only strict follow-up should a complete response after downstaging treatments have been achieved

INTERVENTIONS:
Procedure: Liver transplantation — Once randomized to Group 1, patients will be enlisted for liver transplantation at the recruiting Center. Prioritization is encouraged as a waiting time of more than 8 months could cause patients' drop-out from the study
  Arms: Group 1 - Transplant strategy

SUMMARY:
This clinical trial is aimed at extending the chance of liver transplantation, through downstaging procedures, to patients with hepatocellular carcinoma (HCC) exceeding conventional Milan Criteria.

Those patients that will achieve a sustained tumor response after downstaging will be randomized either to undergo liver transplantation or to proceed with conventional non-transplant treatments.

The aim of the study is to demonstrate unequivocally that liver transplantation may provide a survival benefit, with an acceptable survival rate of at least 60% at 5 years, to patients that demonstrate a radiological and sustained tumor response after downstaging. Noteworthy is that response is chosen rather than stage migration as endpoint of downstaging.

DETAILED DESCRIPTION:
1. Downstaging phase

   Patients that will be considered eligible for the study will undergo downstaging procedures according their stage of disease and to Center's policies. Length and intensity of downstaging will be center specific and not centrally pre-determined, but should be inferior to 18 months. Downstaging procedures will be stopped when, according to the Investigators' judgement, the best possible tumor response has been achieved: at this timepoint a radiological evaluation of tumor response according to modified RECIST (mRECIST) criteria will be performed. Patients that have achieved a Complete or Partial Response (PR or CR) will proceed to Bridging Phase, while those with a Stable or Progressive disease (SD or PD) will drop-out from the study.
2. Bridging phase

   Patients that achieved PR or CR after downstaging will receive systemic therapy with sorafenib for three months. After three months radiological response will be assessed according to mRECIST criteria. If a sustained response will be demonstrated patients will proceed to randomization. PD during bridging phase will cause drop-out from the study.
3. Randomization and study period

Patients will be randomized in a 1:1 ratio, using computer generated list stratified by Center and by compliance to sorafenib treatment (based on whether ≤50% or > 50% of the standard dosage (800 mg/day) has been administered).

1. The experimental group (Group 1 - transplant strategy) will be enlisted for transplantation and will undergo liver transplantation within 8 months unless major medical or oncological contraindications should occur.
2. The control group (Group 2 - non-transplant strategy) will continue with sorafenib until progression. Then they may be treated with either medical or locoregional/surgical therapies according to best practice and Centers' policy, excluding transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patient's age ≥ 18 yrs and ≤ 65 yrs
* Presence of cirrhosis of any etiology
* Child-Pugh class ≤ B7
* ECOG Performance Status ≤ 1
* Diagnosis of HCC either by biopsy or according to AASLD criteria
* HCC exceeding Milan Criteria with a 5-yr estimated survival after transplantation >50% according to the Metroticket calculator (http://www.hcc-olt-metroticket.org/calculator)
* Women of child bearing potential with a negative serum pregnancy test performed before enrolment
* Absence of general contraindications to sorafenib/molecular targeted therapies

Exclusion Criteria:

* Presence of extra-hepatic tumor spread
* Presence of macrovascular invasion
* Sorafenib therapy started > 2 months before enrolment
* Concurrent cancer, distinct from HCC (except cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors)
* Previous history of any cancer, even if curatively treated, < 5 years prior to entry
* Active intra-venous or alcohol abusers
* HIV infection
* History of serious cardiac disease
* Severe pulmonary hypertension not treatable by medical therapy
* Patients with a life expectancy of less than 3 months due to HCC or less than 6 months due to any other disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2011-01; Primary Completion 2015-03-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
For Phase II - Time to Tumoral Event (TTE) | Every 4 months
  TTE after randomization will be calculated as the interval between the randomization date and the date of tumour recurrence for tumor-free patients (either because of liver transplantation or complete response after downstaging procedures) or the date of tumour progression otherwise, with censoring at the date of last contact for event-free patients.
For Phase III - Overall Survival | Every 4 months
  Time form the date of randomization and the date of death, with censoring at the date of last contact for event-free patients

SECONDARY OUTCOMES:
Transplant vs. non transplant strategy cost-benefit analysis | Approx. 1 year after the last patient randomized
  Comparison between the cost/benefit of a downstaging strategy followed by liver transplantation (treatment group) Vs the cost/benefit of convenional therapies (control group), analyzed according to the Quality Adjusted Life Years (QALY) gained in the treatment group
Validation of modified RECIST criteria of radiological response to downstaging treatments | Approx. 8 months after the last patient randomized
  Radiology/pathology correlation on efficacy of downstaging treatments in achieving tumor response, as a basis for possible validation of modified RECIST criteria.
Validation of the Metroticket model for the prognosis of survival after liver transplantation in patients exceeding Milan Criteria | Approx. 1 year after the last patient randomized
  http://www.hcc-olt-metroticket.org/

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Mazzaferro, MD, Principal Investigator — Istituto Nazionale Tumori, Milano
Locations (10):
- Italy (10):
  - Ospedali Riuniti di Bergamo, Bergamo
  - Ospedale Maggiore di Milano Policlinico, Milan
  - Istituto Nazionale Tumori, Milan
  - Azienda Ospedaliera Ospedale Niguarda Ca' Granda, Milan
  - Azienda Ospedaliera Universitaria di Padova, Padua
  - Istituto Mediterraneo per i Trapianti e Terapie ad Alta Specializzazione (ISMETT), Palermo
  - Policlinico Tor Vergata, Roma
  - Ospedale "Lazzaro Spallanzani", Roma
  - Ospedale Umberto Iº Policlinico di Roma, Roma
  - Ospedale Universitario Molinette S. Giovanni Battista di Torino, Torino

REFERENCES:
- [Background] Mazzaferro V, Llovet JM, Miceli R, Bhoori S, Schiavo M, Mariani L, Camerini T, Roayaie S, Schwartz ME, Grazi GL, Adam R, Neuhaus P, Salizzoni M, Bruix J, Forner A, De Carlis L, Cillo U, Burroughs AK, Troisi R, Rossi M, Gerunda GE, Lerut J, Belghiti J, Boin I, Gugenheim J, Rochling F, Van Hoek B, Majno P; Metroticket Investigator Study Group. Predicting survival after liver transplantation in patients with hepatocellular carcinoma beyond the Milan criteria: a retrospective, exploratory analysis. Lancet Oncol. 2009 Jan;10(1):35-43. doi: 10.1016/S1470-2045(08)70284-5. Epub 2008 Dec 4. PMID 19058754
- [Background] Mazzaferro V, Regalia E, Doci R, Andreola S, Pulvirenti A, Bozzetti F, Montalto F, Ammatuna M, Morabito A, Gennari L. Liver transplantation for the treatment of small hepatocellular carcinomas in patients with cirrhosis. N Engl J Med. 1996 Mar 14;334(11):693-9. doi: 10.1056/NEJM199603143341104. PMID 8594428
- [Background] Llovet JM, Di Bisceglie AM, Bruix J, Kramer BS, Lencioni R, Zhu AX, Sherman M, Schwartz M, Lotze M, Talwalkar J, Gores GJ; Panel of Experts in HCC-Design Clinical Trials. Design and endpoints of clinical trials in hepatocellular carcinoma. J Natl Cancer Inst. 2008 May 21;100(10):698-711. doi: 10.1093/jnci/djn134. Epub 2008 May 13. PMID 18477802
- [Background] Lencioni R, Llovet JM. Modified RECIST (mRECIST) assessment for hepatocellular carcinoma. Semin Liver Dis. 2010 Feb;30(1):52-60. doi: 10.1055/s-0030-1247132. Epub 2010 Feb 19. PMID 20175033
- [Derived] Mazzaferro V, Citterio D, Bhoori S, Bongini M, Miceli R, De Carlis L, Colledan M, Salizzoni M, Romagnoli R, Antonelli B, Vivarelli M, Tisone G, Rossi M, Gruttadauria S, Di Sandro S, De Carlis R, Luca MG, De Giorgio M, Mirabella S, Belli L, Fagiuoli S, Martini S, Iavarone M, Svegliati Baroni G, Angelico M, Ginanni Corradini S, Volpes R, Mariani L, Regalia E, Flores M, Droz Dit Busset M, Sposito C. Liver transplantation in hepatocellular carcinoma after tumour downstaging (XXL): a randomised, controlled, phase 2b/3 trial. Lancet Oncol. 2020 Jul;21(7):947-956. doi: 10.1016/S1470-2045(20)30224-2. PMID 32615109
- See also: The system will calculate the 3 and 5 year predicted survival of a given patient with HCC undergoing liver transplantation — http://www.hcc-olt-metroticket.org/